CLINICAL TRIAL: NCT02893566
Title: Effects of A Mi Band Step Challenge on Improving Physical Activity, Sedentary Behavior, and Body Composition in Overweight University Students
Brief Title: Mi Band Step Challenge to Improve Body Composition in Overweight University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Lin, Yun-Ping, Assistant Professor, China Medical University, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 105-2815-C-039-030-B
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Intervention Study; Physical Activity
Keywords: overweight; body mass index; university students; physical activity; sedentary behavior; body composition; Mi Band
MeSH Terms: conditions — Motor Activity; Overweight; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: One group pretest-midtest-posttest design
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mi Band Step Challenge (Experimental)
  Interventions: Behavioral: Mi Band Step Challenge

INTERVENTIONS:
Behavioral: Mi Band Step Challenge

SUMMARY:
This is an eight-month research project using one group pretest-midst-posttest design. This study is based on self-efficacy and self-regulation of Social Cognitive Theory. The investigators will recruit 50 university students with a body mass index of 24 kg/m2 or above at one university campus. Participation is completely voluntary. After pretesting, a 12-week "Mi Band Step Challenge" will be launched immediately. Participants will be assessed with the validated instruments of International Physical Activity Questionnaire (IPAQ)-Taiwan short-form, Sedentary Behavior Questionnaire (SBQ), self-efficacy and self-regulation questionnaires. Mi Band activity trackers will be used to monitor step counts. An ioi 353 body composition analyzer will be used to assess body composition. Data will be analyzed using generalized estimating equation (GEE).

The expected outcomes of this study include: (1) "Mi Band Step Challenge" will be developed based on the theory, which is expected to be effective. If this is true, the intervention can be packaged and applied at different types of colleges and universities with overweight students. (2) "Mi Band Step Challenge" has the potential to be used for the reference of the healthy weight - physical activity, which is embedded in the School Health Promotion Program executed by the Ministry of Education. (3) The result of this study can serve as an example for the promotion of evidence-based health care.

ELIGIBILITY:
Inclusion Criteria:

* University students with a body mass index of 24 kg/m2 or above at one university campus.
* No physical limitations that would prevent them from performing physical activity.
* Not currently pregnant women.
* Having a smart phone that would allow them to connect to a Mi Band.

Exclusion Criteria:

* The university student who expects to be absent for more than 2 weeks or expects a suspension or transferring to another school during the implementation of the intervention.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Weight | Change from baseline weight at 6 weeks and 12 weeks
  Weight was measured by ioi 353 body composition analyzer (Jawon Medical)
Waist circumference (WC) | Change from baseline waist circumference at 6 weeks and 12 weeks
  Waist circumference (nearest 0.1 cm) was measured in duplicate with a non-expandable tape at the midpoint between the lowest rib and the iliac crest. A third measurement was taken if the first two differed by 1 cm.
Soft lean mass (SLM) | Change from baseline soft lean mass at 6 weeks and 12 weeks
  Soft lean mass was measured by ioi 353 body composition analyzer (Jawon Medical)
Mass of body fat (MBF) | Change from baseline mass of body fat at 6 weeks and 12 weeks
  Mass of body fat was measured by ioi 353 body composition analyzer (Jawon Medical)
Percent body fat (PBF) | Change from baseline percent body fat at 6 weeks and 12 weeks
  Percent body fat was measured by ioi 353 body composition analyzer (Jawon Medical)
Body mass index (BMI) | Change from baseline body mass index at 6 weeks and 12 weeks
  Body mass index was computed as average weight (kg)/average height (m2)
Waist to hip ratio (WHR) | Change from baseline waist to hip ratio at 6 weeks and 12 weeks
  Waist to hip ratio was measured by ioi 353 body composition analyzer (Jawon Medical)

SECONDARY OUTCOMES:
Physical activity | Change from baseline physical activity at 6 weeks and 12 weeks
  Physical activity was assessed by International Physical Activity Questionnaire (Taiwan) short-form (IPAQ-SF)
Sedentary behavior | Change from baseline sedentary behavior at 6 weeks and 12 weeks
  Sedentary behavior was assessed by Rosenberg's Sedentary Behavior Questionnaire (SBQ)
Daily steps | Change from baseline daily steps at 6 weeks and 12 weeks
  Daily steps was assessed by Mi Band (Xiaomi Inc.)

OTHER OUTCOMES:
Self-regulation questionnaire | Change from baseline self-regulation at 6 weeks and 12 weeks
Self-efficacy for physical activity questionnaire | Change from baseline self-efficacy for physical activity at 6 weeks and 12 weeks
Self-efficacy for reducing sedentary behavior questionnaire | Change from baseline self-efficacy for reducing sedentary behavior at 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Ping Lin, PhD, Principal Investigator — China Medical University, China